CLINICAL TRIAL: NCT05416879
Title: Lifestyle Behaviours of Women Newly Diagnosed With Heart Failure: A Quantitative and Qualitative Approach
Brief Title: Lifestyle Behaviours of Women Newly Diagnosed With Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 308745
Record Dates: First submitted 2022-05-12; First posted 2022-06-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Women newly diagnosed with heart failure
  Interventions: Device: Actigraph GT3X+BT

INTERVENTIONS:
Device: Actigraph GT3X+BT — 7 day monitoring of physical activity, sedentary behaviour and sleep using the Actigraph GT3X+BT

SUMMARY:
Heart Failure occurs when the heart's ability to pump blood is reduced. Heart failure can lead to symptoms of breathlessness, fatigue and ankle swelling, and result in health complications including damage to other organs (e.g. kidneys), reduced function and quality of life. Although the symptoms of heart failure are similar for men and women, there are sex differences. Lifestyle behaviours such as physical activity are important modifiable risk factor for heart failure. Women continue to be underrepresented in heart failure studies and treatment guidelines are male-derived due to these disparities in recruitment. The purpose of the present study is to evaluate the physical activity levels, sedentary behaviour, sleep and quality of life and understand the barriers and facilitators to these lifestyle behaviours in women newly diagnosed with heart failure.

DETAILED DESCRIPTION:
Background: Heart failure is a condition in which the heart has a reduced function to pump blood during exertion and often at rest. Although the symptoms for heart failure are similar for men and women, there are sex differences in the heart failure etiologies. The incidence of heart failure is greater in men versus women, especially in the younger age groups (45-54 years). However, it has been reported from 79 years old, women have a greater prevalence than men. This is associated with the age at diagnosis being 5 years older for women compared to men (79.6 vs. 74.8 years). Men are more likely to present with heart failure with reduced ejection fraction (HFrEF) whereas women are twice as likely to present with heart failure with preserved ejection fraction (HFpEF). Given their more complex medical profile, men have significantly higher healthcare costs versus women during the first year after diagnosis. The global COVID-19 pandemic has resulted in services and care for patients with heart failure being significantly affected. Our recent review highlighted that patients are continuing to avoid urgent care, which may result in advanced manifestations of cardiac dysfunction and worse prognosis.

Physical activity is an important modifiable risk factor in patients with chronic heart failure and is known to improve function and quality of life (QoL). Although several studies report physical activity in patients with chronic heart failure, it appears that no study has evaluated physical activity in women at the time of diagnosis of heart failure and evaluated these lifestyle behaviours by understanding the barriers and facilitators. Women are underrepresented in heart failure studies and treatment guidelines are male-derived due to these disparities in recruitment. Our research will directly address this by evaluating the physical activity levels, sedentary behaviour, sleep and QoL of women newly diagnosed with heart failure and understand the barriers and facilitators to these lifestyle behaviours at the time of diagnosis.

Aim and Objectives: The aim of the project is to provide evidence for the current lifestyle behaviors of women newly diagnosed with heart failure. The aim will be achieved through the following three objective: (1) assess the physical activity levels, sedentary behavior and sleep of women newly diagnosed with heart failure using objective assessment (2) evaluate the quality of life of women newly diagnosed with heart failure and (3) understand the barriers and facilitators of these lifestyle behaviors of women at the time of their heart failure diagnosis.

Methods/Design: Study Design: A prospective, single-centre, pilot study design will evaluate physical activity, sedentary behaviour, sleep and QoL of women newly diagnosed with heart failure who have been referred to secondary care for specialist review and have attended a heart failure diagnostic clinic at the Royal Victoria Infirmary, Newcastle-upon-Tyne.

Recruitment procedures: Participants will be identified from the Heart Failure Diagnostic Clinics run by Drs MacGowan and Bailey who are part of the research study team and play a vital role in participant recruitment. An information sheet will be given to all patients (women only) after they have received their diagnosis at the diagnostic clinic appointment. A member of the research study team will attend the Heart Failure Diagnostic Clinics to provide a participant information sheet to eligible patients. The research study team will have an honorary contract with the Newcastle upon Tyne Hospital and sufficient level of competence and permission to assess patients' medical records using computerised system in place. The patient will be given at least 48 hours to read through the participant information sheet. A member of the research team will contact the patient via telephone call to see if they are happy to participate in the study. Research will seek informed and voluntary consent from the participant. A consent form will be attached to the participant information sheet for the patient to complete and return to the research study team via a pre-paid envelope. Consent forms will be signed by the participant and countersigned by a member of the research study team.

Part 1: Quantitative Work Package: As part of the standard care and practice in at the Royal Victoria Infirmary (RVI), the following investigations will be performed by specialist NHS staff members:

1. Echocardiography for assessment of cardiac structure and function using non-invasive Doppler ultrasound (30 min).
2. Medical history review, physical examination and interpretation of echocardiography results by a consultant cardiologist, who is also part of the research team, confirming or ruling out heart failure diagnosis (30 min).

Wrist monitor and questionnaires: A total of 40 newly diagnosed heart failure patients will be recruited to the study. Once the research study team has received the participant's postal consent form, a study pack will be posted to the participant, which will include: a wrist monitor, a set of instructions, two validated questionnaires and a pre-paid envelope to return the wrist monitor and questionnaires. By completing this part of the study remotely, the patient will avoid making an additional visit to the hospital at the time of diagnosis.

The participant will be asked to wear the wrist monitor (Actigraph GT3X+BT) to capture habitual 7-day physical activity, sedentary behaviour and sleep on one occasion. A set of instructions will be posted with the wrist monitor and the research study team telephone contact details will be provided. A follow-up telephone call will be made to the participant to ensure they have received all the information and are happy to complete the questionnaires and 7 day monitoring.

The two validated questionnaires are the Minnesota Living with Heart Failure (MLHF) Questionnaire and the SF-36 and the participant will be asked to complete these prior to completing the 7-day monitoring.

The participant will receive a small padded pre-paid envelope to post the wrist monitor and questionnaires to the research study team at the end of the 7 days monitoring. The wrist monitor data will be processed using the ActiLife software.

The MLHF and SF-36 questionnaires will be posted to the participant at 3 months post-diagnosis to assess any short-term changes in QoL. A pre-paid envelope will be provided to the participant to return the questionnaires to the research study team.

Part 2: Qualitative Work Package: In parallel to the quantitative work package, it is important to clarify what are the barriers and facilitators to these important lifestyle behaviours, i.e. physical activity, sedentary behaviours, sleep and QoL at the time of diagnosis for women. The aim of this work package is to understand what lifestyle behaviours participants currently engage in at the time of diagnosis and how their diagnosis may affect their future lifestyle choices.

One optional semi-structured interviews will be conducted with the participants who provide consent to participate in this part of the study (n=15 or until saturation in findings) once they have completed the quantitative work package. Participants may choose to opt out from this part of the study and this option will be included in the consent form. An interview specific topic guide has been developed on the barriers and facilitators to physical activity, sedentary behaviours, sleep and QoL. Data from the semi-structured interviews will be analysed thematically using an inductive approach. All interviews will be transcribed verbatim. The interviews will be conducted remotely and participants will be given the option to use the zoom platform or receive a telephone call. If the participant becomes distressed or upset from completing the interview (and/or the questionnaires) then the investigators have requested they contact the research study team who will initiate referral to our clinical psychology department at the Freeman Hospital or Royal Victoria Infirmary, Newcastle upon Tyne.

Sample size and statistical analysis: The quantitative work package will produce pilot study findings and a recruitment target of 40 patients was chosen, which will adhere to methodological standards for pilot studies. Descriptive statistics of the data variables (physical activity levels, sedentary behaviour, sleep and QoL) will be analysed and compared to age and sex-matched healthy controls. Data (natriuretic peptides (NTproBNP) and left ventricular ejection fraction (LVEF)) from patient's medical records will be exported.

The qualitative work package will involve a purposely selected sample of women with a new diagnosis of heart failure (n=15). This is exploratory work, therefore, an inductive approach to analysis will be made and data saturation of themes will be determined at the analysis stage. Two independent investigators in the research study team will code and extract segments of the data to identify key themes. Inclusion of supporting quotes from each of the themes will be included in the write up and publication.

Funding: This study has received funding from the Wellcome Trust ISSF scheme.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with a new diagnosis of heart failure after referral to the RVI Heart Failure Diagnostic Clinic;
* Able to walk and perform activities of daily living independently;
* New York Heart Association functional class II-IV;
* Willingness to undertake physical activity monitoring;
* Willingness to participate in a semi-structured interview (this is optional and the participant will be able to participate in the study if they choose not to take part in the interview);
* Ability to read, write and converse in English without the support of an interpreter;
* Able to provide written informed consent.

Exclusion Criteria:

* Male;
* Already diagnosed with heart failure;
* Presented with severe symptoms requiring urgent assessment and stabilisation (e.g. breathless at rest, hypotension, confusion);
* Major co-morbidity or other alternative diagnoses of no obvious acute and self-limiting cause (e.g. malignancy, severe respiratory disease, mental health problem);
* Severe physical disability preventing them to function independently;
* Clinically unstable with recent changes in medication;
* Unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women newly diagnosed with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of steps per day during a 7-day monitoring period | 7-day at the time of diagnosis
  7-day objective assessment using Actigraph GT3X+BT accelerometry at the time of diagnosis
Intensity of physical activity (light physical activity, measured in minutes per day) during a 7-day monitoring period | 7-day at the time of diagnosis
  7-day objective assessment using Actigraph GT3X+BT accelerometry at the time of diagnosis
Intensity of physical activity (moderate physical activity, measured in minutes per day) during a 7-day monitoring period | 7-day at the time of diagnosis
  7-day objective assessment using Actigraph GT3X+BT accelerometry at the time of diagnosis
Intensity of physical activity (vigorous physical activity, measured in minutes per day) during a 7-day monitoring period | 7-day at the time of diagnosis
  7-day objective assessment using Actigraph GT3X+BT accelerometry at the time of diagnosis
Time spent sedentary (measured in minutes per day) during a 7-day monitoring period | 7-day at the time of diagnosis
  7-day objective assessment using Actigraph GT3X+BT accelerometry at the time of diagnosis
Sleep duration (measured in minutes per day) during a 7-day monitoring period | 7-day at the time of diagnosis
  7-day objective assessment using Actigraph GT3X+BT accelerometry at the time of diagnosis
Change in Baseline Minnesota Living with Heart Failure Questionnaire at 3 months | 3 months
  A 21-item questionnaire. A 5-point Likert scale used for each question. The questions are summed and the minimum and maximum values are 0-105. A higher score represents a worse health-related quality of life.
Change in Baseline 36-Item Short Form Survey Instrument at 3 months | 3 months
  A 36-item survey, which includes eight health concepts (physical functioning (10 items), role limitations due to physical health (4 items), role limitations due to emotional problems (3 items), energy/fatigue (4 items), emotional well-being (5 items), social functioning (2 items), pain (2 items) and general health (5 items). Each item is scored 0-100. A higher score represents a better health-related quality of life.
Patient's perceptions of physical activity, sedentary behaviour and quality of life | 60 minutes
  A semi-structured interview will explore the barriers and opportunities of past, present and future physical activity, sedentary behaviour and quality of life at the time of diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data archive and sharing Research data that supports publications and unpublished data of value at project end will be archived with supporting documentation in data.ncl (https://data.ncl.ac.uk/), Newcastle's Research Data Repository. The datasets will be made public under a Creative Commons licence to ensure credit is given when the data is reused and access provided for at least ten years. Data deposited will also be assigned a persistent identifier (i.e. DOI) that can be included in project outputs, including publications, to detail how and where the data can be accessed. At this stage all study identification numbers will be removed and all data will be anonymised before being archived and shared through the repository. Where there is a risk to data being re-identified the dataset will be archived to make the record findable but access will be controlled and dependent on the future use of the data in question.
Time Frame: 5 years

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Eisenberg E, Di Palo KE, Pina IL. Sex differences in heart failure. Clin Cardiol. 2018 Feb;41(2):211-216. doi: 10.1002/clc.22917. Epub 2018 Feb 27. PMID 29485677
- [Background] Conrad N, Judge A, Tran J, Mohseni H, Hedgecott D, Crespillo AP, Allison M, Hemingway H, Cleland JG, McMurray JJV, Rahimi K. Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals. Lancet. 2018 Feb 10;391(10120):572-580. doi: 10.1016/S0140-6736(17)32520-5. Epub 2017 Nov 21. PMID 29174292
- [Background] Shin JJ, Hamad E, Murthy S, Pina IL. Heart failure in women. Clin Cardiol. 2012 Mar;35(3):172-7. doi: 10.1002/clc.21973. PMID 22389122
- [Background] Taylor CJ, Ordonez-Mena JM, Jones NR, Roalfe AK, Lay-Flurrie S, Marshall T, Hobbs FDR. National trends in heart failure mortality in men and women, United Kingdom, 2000-2017. Eur J Heart Fail. 2021 Jan;23(1):3-12. doi: 10.1002/ejhf.1996. Epub 2020 Sep 23. PMID 32892471
- [Background] Cremers, H., et al. Gender differences in Heart Failure; Data on Outcomes and Costs. ESC European Society of Cardiology, 2020
- [Background] Charman SJ, Velicki L, Okwose NC, Harwood A, McGregor G, Ristic A, Banerjee P, Seferovic PM, MacGowan GA, Jakovljevic DG. Insights into heart failure hospitalizations, management, and services during and beyond COVID-19. ESC Heart Fail. 2021 Feb;8(1):175-182. doi: 10.1002/ehf2.13061. Epub 2020 Nov 24. PMID 33232587
- [Background] Cattadori G, Segurini C, Picozzi A, Padeletti L, Anza C. Exercise and heart failure: an update. ESC Heart Fail. 2018 Apr;5(2):222-232. doi: 10.1002/ehf2.12225. Epub 2017 Dec 13. PMID 29235244
- [Background] Jakovljevic DG, McDiarmid A, Hallsworth K, Seferovic PM, Ninkovic VM, Parry G, Schueler S, Trenell MI, MacGowan GA. Effect of left ventricular assist device implantation and heart transplantation on habitual physical activity and quality of life. Am J Cardiol. 2014 Jul 1;114(1):88-93. doi: 10.1016/j.amjcard.2014.04.008. Epub 2014 Apr 18. PMID 24925802
- [Background] Okwose NC, Avery L, O'Brien N, Cassidy S, Charman SJ, Bailey K, Velicki L, Olivotto I, Brennan P, MacGowan GA, Jakovljevic DG. Acceptability, Feasibility and Preliminary Evaluation of a Novel, Personalised, Home-Based Physical Activity Intervention for Chronic Heart Failure (Active-at-Home-HF): a Pilot Study. Sports Med Open. 2019 Nov 27;5(1):45. doi: 10.1186/s40798-019-0216-x. PMID 31776701
- [Background] Riegel B, Moser DK, Glaser D, Carlson B, Deaton C, Armola R, Sethares K, Shively M, Evangelista L, Albert N. The Minnesota Living With Heart Failure Questionnaire: sensitivity to differences and responsiveness to intervention intensity in a clinical population. Nurs Res. 2002 Jul-Aug;51(4):209-18. doi: 10.1097/00006199-200207000-00001. PMID 12131233
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Virginia Braun & Victoria Clarke (2006) Using thematic analysis in psychology, Qualitative Research in Psychology, 3:2, 77-101, DOI: 10.1191/1478088706qp063oa
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Saunders B, Sim J, Kingstone T, Baker S, Waterfield J, Bartlam B, Burroughs H, Jinks C. Saturation in qualitative research: exploring its conceptualization and operationalization. Qual Quant. 2018;52(4):1893-1907. doi: 10.1007/s11135-017-0574-8. Epub 2017 Sep 14. PMID 29937585

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT05416879/Prot_SAP_000.pdf